CLINICAL TRIAL: NCT05498350
Title: Randomized Trial Comparing Early "Trigger" Versus Delayed "Trigger" Timing in Cycles of Controlled Ovarian Stimulation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fertility Center of Las Vegas (Industry)
Responsible Party: Principal Investigator, Bruce Shapiro M.D., Medical Director, Fertility Center of Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCLV-2022-1
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Trigger (Experimental)
  Interventions: Procedure: Ovulatory trigger timing
- Delayed trigger (Experimental)
  Interventions: Procedure: Ovulatory trigger timing

INTERVENTIONS:
Procedure: Ovulatory trigger timing — Timing of medication to induce final oocyte maturation

SUMMARY:
This randomized trial will compare the efficacy of two different times of administration of medications for final oocyte maturation, commonly called a "trigger", in cycles of controlled ovarian stimulation (COS) for cycles in which all embryos will be cryopreserved ("freeze-all cycles").

DETAILED DESCRIPTION:
This randomized trial will compare the efficacy of two different times of administration of medications for final oocyte maturation, commonly called a "trigger", in cycles of controlled ovarian stimulation (COS) for cycles in which all embryos will be cryopreserved ("freeze-all cycles").

1. The early trigger timing will be based on sonographic observation of at least three follicles reaching at least 17mm in diameter.
2. The delayed trigger timing will be based on at least three follicles reaching at least 22mm in diameter.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female at least 18 years of age and less than 35 years of age intending to undergo ovarian stimulation for a cycle of IVF with all embryos to be frozen that attain the blastocyst stage.
2. Anticipated at least normal ovarian response evidenced by at least 8 antral follicles observed on ultrasound or a serum level of at least 1.5 ng/ml AMH.
3. Ability read and understand English sufficiently to obtain informed consent.
4. Patients with prior IVF cycles are allowed, but no patient can undergo more than one cycle with oocyte collection under this study.

Exclusion Criteria:

1. Any cycle type that would preclude immediate culture to blastocyst stage (e.g. oocyte banking).
2. Any condition that, in the opinion of the physician or principal investigator, would place the patient at undue risk under this protocol or would otherwise make the protocol inappropriate for that subject.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Good-quality blastocysts | Within 7 days of oocyte retrieval
  Number of blastocysts with A or B morphological grade.
Delayed blastocyst formation | Within 7 days of oocyte retrieval
  Proportion of good-quality of blastocysts that formed after day 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility center of Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No